CLINICAL TRIAL: NCT00634257
Title: A Preliminary Study of Spirituality/Religiosity, Symptom Distress and Quality of Life Among Palliative Care Patients and Their Primary Caregivers
Brief Title: Spirituality/Religiosity in Patients and Caregivers
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0678; NCI-2011-02785 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-02-25; First posted 2008-03-12 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Advanced Cancer; Solid Tumors
Keywords: Advanced Cancer; Solid Tumors; Spirituality; Religiosity; Symptom Distress; Quality of Life; Caregivers; Questionnaire; Survey
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with advanced cancer receiving palliative care.
  Interventions: Behavioral: Questionnaires
- Caregivers: Primary caregivers of Patients with advanced cancer receiving palliative care.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Nine questionnaires taking about 40 minutes to complete.
  Other Names: Survey

SUMMARY:
Primary Objective:

-To examine the association between self-rated spirituality/religiosity and coping strategies (Brief RCOPE, Brief COPE, SBI-15R) among palliative care patients.

Secondary Objectives:

* To examine the associations between self-rated spirituality/religiosity and physical (ESAS) and psychological symptom reports (HADS), and quality of life (FACIT-sp) among palliative care patients.
* To examine the association between patient's self-reported spirituality/religiosity, and primary caregiver distress (HADS, PSQI, CQLS-C, caregiver self-assessment questionnaire, FACIT-sp).
* To determine the frequency (self-rated spiritual pain scale when score is more or equal than 1 in the scale 0 to 10) and intensity of self-rated spiritual pain in the palliative care setting and to explore the association between spiritual pain, and negative religious coping (Brief RCOPE), physical (ESAS) and psychological symptoms (HADS), and primary caregiver distress (CQLS-C, caregiver self-assessment questionnaire).
* To examine the association between primary caregivers' spirituality/religiosity (Appendix H, first question), religious coping strategies (Brief-RCOPE) and psychological and family/caregiver distress (HADS, PSQI, CQLS-C, caregiver self-assessment questionnaire), and caregivers' spiritual pain (Appendix F, second question).

DETAILED DESCRIPTION:
Questionnaires:

If you are found to be eligible to take part in this study and you agree to take part, you will complete 9 questionnaires.

The first 2 questionnaires ask about your demographic information (such as your education level and age) and the symptoms of cancer you may be experiencing.

The 6 other questionnaires ask questions about several subjects. You will be asked about your religious/spiritual beliefs, such as your way of coping with cancer and whether you have focused on religion/spirituality or other strategies in order to stop worrying. You will also be asked whether you feel religious/spiritual beliefs are important in your everyday life, how hopeful you may feel, and the level of spiritual pain you may feel. (Some people experience spiritual pain as a deep pain in the "soul" or "being" that is not physical pain.)

The last questionnaire asks about any symptoms of anxiety or depression you may feel. In total, these questionnaires should take about 40 minutes to complete.

Length of Study Participation:

After completing the questionnaires, your participation in this study will be over.

This is an investigational study. Up to 100 patients and 100 caregivers will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. (Patients) Advanced cancer patients seen in palliative care outpatient clinic and palliative care mobile team and inpatient unit at M.D. Anderson Cancer Center
2. (Patients) Patients aged 18 years or over
3. (Patients) Karnofsky performance status score of more than 40 at time of inclusion into study. (Patients with Karnofsky score less than 40 may not be able to complete the measures).
4. (Patients) Able to provide informed consent and comply with study procedures
5. (Caregivers) Spouse, first degree relative, or other person designated by the patient as providing direct assistance to the patient in his/her activities of daily living
6. (Caregivers) Having the patient's consent to be contacted.
7. (Caregivers) Caregiver is 18 years or over
8. (Caregivers) Able to provide informed consent and comply with study procedures
9. (Patients) only English-speaking, as determined by their ability to understand the informed consent and the assessment tools.
10. (Caregivers) only English-speaking, as determined by their ability to understand the informed consent and the assessment tools.
11. (Patients) Normal cognitive status as determined by the interviewer based on the ability to understand the nature of the study and consent process.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer receiving palliative care and their primary caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2008-02-22 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Association between self-rated spirituality/religiosity and coping strategies | Questionnaires completed by patient/caregiver at second consult visit, estimate 40 minutes to finish forms.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org